CLINICAL TRIAL: NCT00815035
Title: Oral Immunotherapy for Peanut Allergy- Peanut Oral Immunotherapy (PnOIT3)
Brief Title: Oral Immunotherapy (OIT) for Peanut Allergy
Acronym: PnOIT3
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: 11-2315
Record Dates: First submitted 2008-12-26; First posted 2008-12-29 (Estimated); Results first posted 2017-05-15 (Actual); Last update posted 2018-03-01 (Actual); Status verified 2017-07

CONDITIONS: Peanut Hypersensitivity
Keywords: Peanut Allergy
MeSH Terms: conditions — Peanut Hypersensitivity

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Peanut OIT (Active Comparator): Subjects randomized to receive active treatment with peanut protein flour.
  Interventions: Drug: Peanut OIT
- Placebo (Placebo Comparator): Subjects randomized to receive placebo in the form of oat flour.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Peanut OIT — Peanut flour that is orally ingested in a graded fashion.
  Other Names: Peanut flour
  Arms: Peanut OIT
Drug: Placebo — Oat flour used as a placebo that is orally ingested a graded fashion
  Other Names: Oat flour
  Arms: Placebo

SUMMARY:
Peanut allergy is known to cause severe anaphylactic reactions.The goal of this proposal is to produce a new treatment that would benefit subjects who have peanut allergy by lowering the risk of anaphylactic reactions (desensitization), and changing the peanut-specific immune response in subjects who have peanut allergy (tolerance).

DETAILED DESCRIPTION:
Peanut allergy is known to cause severe anaphylactic reactions. Compared with other food allergies it tends to be more persistent and also its prevalence seems to be rising. Currently there is no proven treatment other than strict avoidance. We are attempting to decrease the risk of anaphylaxis on accidental ingestion by desensitizing subjects to peanut using peanut oral immunotherapy (OIT). We are also studying the effect of peanut OIT on the peanut specific immune response to determine if tolerance to peanut protein will develop. Children ages one to six years of age with peanut allergy will be randomized to peanut OIT or placebo (active subjects). Thirty subjects will also be recruited as controls. These subjects will not receive any peanut or placebo but only have skin prick testing and lab work in addition to a history and physical exam. Active subjects will undergo a modified rush immunotherapy on the first day and then increase the doses at least every two weeks up to a maintenance dose of 4 grams (equivalent to about 13 peanuts). Doses will be taken daily at home except for dose increases which will be done on the research unit. Outcome variables of interest include response to double-blind placebo controlled food challenge, skin prick testing, peanut specific IgE, and adverse events. These results will be compared between the start and end of peanut OIT using appropriate statistical analysis.

ELIGIBILITY:
Inclusion Criteria:

* Age 1- 6 years all of either sex, any race, any ethnicity at the time of the initial visit
* The presence of IgE specific to peanuts (a positive skin prick test to peanuts (diameter of wheal >3.0 mm) and a positive in vitro IgE [CAP-FEIA] > 7 kUA/L
* A history of significant clinical symptoms occurring within 60 minutes after ingesting peanuts
* Provide signed informed consent

Exclusion Criteria:

* History of severe anaphylaxis to peanut as defined by hypoxia, hypotension, or neurological compromise (Cyanosis or oxygen saturation < 92% at any stage, hypotension, confusion, collapse, loss of consciousness; or incontinence)
* Currently participating in a study using an investigational new drug
* Participation in any interventional study for the treatment of food allergy in the past 12 months
* Subjects with a known wheat food allergy will be excluded because of cross contamination of oat with wheat
* Poor control or persistent activation of atopic dermatitis
* Moderate to severe persistent asthma
* Currently being treated with greater than medium daily doses of inhaled corticosteroids, as defined by the National Heart Lung and Blood Institute (NHLBI) guidelines
* Inability to discontinue antihistamines for skin testing and oral food challenges (OFCs)

Ages: 1 Year to 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 16 (Actual)
Dates: Start 2009-04; Primary Completion 2016-12-12 (Actual); Study Completion 2016-12-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Wesley Burks, MD, Principal Investigator — University of North Carolina
Locations (1):
- University of North Carolina, Chapel Hill, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Patriarca G, Nucera E, Roncallo C, Pollastrini E, Bartolozzi F, De Pasquale T, Buonomo A, Gasbarrini G, Di Campli C, Schiavino D. Oral desensitizing treatment in food allergy: clinical and immunological results. Aliment Pharmacol Ther. 2003 Feb;17(3):459-65. doi: 10.1046/j.1365-2036.2003.01468.x. PMID 12562461
- [Background] Buchanan AD, Green TD, Jones SM, Scurlock AM, Christie L, Althage KA, Steele PH, Pons L, Helm RM, Lee LA, Burks AW. Egg oral immunotherapy in nonanaphylactic children with egg allergy. J Allergy Clin Immunol. 2007 Jan;119(1):199-205. doi: 10.1016/j.jaci.2006.09.016. Epub 2006 Oct 27. PMID 17208602

RESULTS

PARTICIPANT FLOW:
Groups:
- Blinded Phase-Peanut OIT: Subjects randomized over the initial 44+ weeks to receive active treatment with peanut OIT.
  Peanut OIT: Peanut flour that is orally ingested in a graded fashion.
- Blinded Phase-Placebo: Subjects randomized over the first 44+ weeks to receive placebo in the form of oat flour.
  Placebo: Oat flour used as a placebo that is orally ingested a graded fashion
- Open Label Phase-Peanut OIT: Subjects receiving open-label peanut OIT treatment after unblinding through the end of study.
  Peanut OIT: Peanut flour that is orally ingested in a graded fashion.
Period: Blinded Phase
Arm/Group | Blinded Phase-Peanut OIT | Blinded Phase-Placebo | Open Label Phase-Peanut OIT
Started | 10 | 6 | 0
Completed | 9 | 6 | 0
Not Completed | 1 | 0 | 0
Period: Open Label Extension Phase
Arm/Group | Blinded Phase-Peanut OIT | Blinded Phase-Placebo | Open Label Phase-Peanut OIT
Started | 0 (After unblinding, subjects completing the blinded phase moved to the open-label phase of the study) | 0 (After unblinding, subjects completing the blinded phase moved to the open-label phase of the study) | 15 (After unblinding, subjects completing the blinded phase moved to the open-label phase of the study)
Completed | 0 | 0 | 9
Not Completed | 0 | 0 | 6

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Blinded Phase-Peanut OIT | Blinded Phase-Placebo | Total
Number analyzed (Participants) | 10 | 6 | 16
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 10 | 6 | 16
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Full Range); unit: years] | 5.1 [3.8 to 6.9] | 4.8 [3.6 to 6.9] | 5.0 [3.6 to 6.9]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 4 | 10
  Male | 4 | 2 | 6
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 10 | 6 | 16
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 0 | 1
  White | 8 | 4 | 12
  More than one race | 1 | 2 | 3
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 10 | 6 | 16

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Subjects Achieving Tolerance as Defined by a Negative DBPCFC 4 Weeks After Discontinuation of Peanut OIT Therapy.
Description: Upon completion of 60 months of peanut OIT treatment, subjects discontinued peanut OIT for 4 weeks. The primary clinical efficacy outcome of the study was the percentage of peanut allergic subjects who completed a 5 gm peanut protein double-blind placebo controlled food challenge (DBPCPFC) without developing symptoms 4 weeks after discontinuing peanut OIT.
Time Frame: 61 months for those randomized to active treatment and 73 months for those randomized to placebo for the initial 12 months of therapy
Population: Subjects completing 60 months of OIT treatment, then passing the DBPCFC on the last day of treatment, then completing the DBPCFC after 1 month off of treatment were analyzed.
Measure: Number; unit: percentage of participants
Arm/Group | Open Label Phase-Peanut OIT
Number analyzed (Participants) | 9
percentage of participants | 89

2. Secondary Outcome: The Percentage of Subjects Achieving Full Desensitization as Defined by a Negative DBPCFC After 60 Months of Peanut OIT Therapy.
Description: Upon completion of 60 months of peanut OIT treatment, subjects underwent a double-blind placebo controlled food challenge (DBPCPFC) to assess desensitization. The secondary clinical efficacy outcome of the study was the percentage of peanut allergic subjects who completed a 5 gm peanut protein double-blind placebo controlled food challenge (DBPCPFC) without developing symptoms after completing peanut OIT therapy.
Time Frame: 60 months for those randomized to active treatment and 72 months for those randomized to placebo for the initial 12 months of therapy
Population: Subjects completing 60 months of OIT treatment and completing the DBPCFC on the last day of treatment were analyzed.
Measure: Number; unit: percentage of participants
Arm/Group | Open Label Phase-Peanut OIT
Number analyzed (Participants) | 9
percentage of participants | 100

3. Secondary Outcome: The Percentage of Subjects Who Tolerated the Initial-day Escalation to 6 mg of Peanut
Description: The first day of peanut OIT dosing involved multiple increasing doses of peanut flour in what was called an initial escalation day up to a maximum dose of 6 mg of peanut protein. The secondary outcome measure assessed the percentage of subjects were successfully able to reach this 6 mg dose.
Time Frame: first day of peanut OIT dosing
Population: Open label phase includes subjects initially randomized to placebo and then subsequently crossed over to open label treatment. Subjects initially randomized to Peanut OIT maintained their dose and did not repeat this 6 mg initial-day escalation.
Measure: Number; unit: percentage of participants
Arm/Group | Blinded Phase-Peanut OIT | Blinded Phase-Placebo | Open Label Phase-Peanut OIT
Number analyzed (Participants) | 10 | 6 | 6
percentage of participants | 90 | 100 | 100

4. Secondary Outcome: The Percentage of Subjects Who Are Successfully Able to Escalate up to the 4000 mg Maximum Maintenance Dose of Peanut Protein OIT During the 60 Month Desensitization Phase of the Study
Description: During the desensitization phase of the study, subjects under go an initial day escalation up to a maximum of 6 mg of peanut protein. They then undergo biweekly dose escalation over approximately 10 months up to a maximum dose of 4000 mg of peanut protein. This outcome reports the percentage of subjects that achieve this.
Time Frame: approximately 40 weeks (10 months)
Population: Open label phase includes subjects initially randomized to placebo and then subsequently crossed over to open label treatment. Subjects initially randomized to Peanut OIT maintained their dose and did not re-escalate for the purposes of this outcome.
Measure: Number; unit: percentage of patients
Arm/Group | Blinded Phase-Peanut OIT | Blinded Phase-Placebo | Open Label Phase-Peanut OIT
Number analyzed (Participants) | 10 | 6 | 6
percentage of patients | 90 | 100 | 66.7

5. Secondary Outcome: Incidence of All Serious Adverse Events During the Study
Description: All serious adverse events during the blinded and open-label phases of the study were recorded and reported as a safety outcome.
Time Frame: 61 months for those randomized to active peanut OIT and 73 months for those randomized to placebo for the initial 12 months of the study.
Population: The initial 10-11 months of the study were blinded. After unblinding, subjects completing the blinded phase continued on open label peanut OIT for the duration of the study.
Measure: Number; unit: number of discrete SAE events
Arm/Group | Blinded Phase-Peanut OIT | Blinded Phase-Placebo | Open Label Phase-Peanut OIT
Number analyzed (Participants) | 10 | 6 | 15
number of discrete SAE events | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Adverse events were collected over the initial 44+ weeks of blinded therapy and then over the 60 month duration of the open-label phase of the study.
Arm/Group | Blinded Phase-Peanut OIT | Blinded Phase-Placebo | Open Label Phase-Peanut OIT
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/6 | 0/15
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/6 | 0/15
Other Adverse Events (participants affected / at risk) | 10/10 | 4/6 | 15/15
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Blinded Phase-Peanut OIT (N=10) | Blinded Phase-Placebo (N=6) | Open Label Phase-Peanut OIT (N=15)
Vomiting (Gastrointestinal disorders) | 9 | 2 | 5
Diarrhea (Gastrointestinal disorders) | 2 | 2 | 3
Erythematous rash (Skin and subcutaneous tissue disorders) | 6 | 1 | 5
Rhinorrhea (Respiratory, thoracic and mediastinal disorders) | 3 | 1 | 4
Wheezing (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 3
Oropharyngeal itching (Skin and subcutaneous tissue disorders) | 9 | 2 | 7
Sneezing (Respiratory, thoracic and mediastinal disorders) | 4 | 2 | 4
Coughing (Respiratory, thoracic and mediastinal disorders) | 6 | 3 | 6
Itchy nose (Skin and subcutaneous tissue disorders) | 3 | 0 | 2
Skin itch (Skin and subcutaneous tissue disorders) | 5 | 2 | 6
Lip or eye swelling (Skin and subcutaneous tissue disorders) | 2 | 1 | 5
Eye itch (Eye disorders) | 1 | 0 | 3
Eye tearing (Eye disorders) | 1 | 0 | 1
Hives (Skin and subcutaneous tissue disorders) | 3 | 2 | 6
Abdominal pain (Gastrointestinal disorders) | 9 | 2 | 11
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No